CLINICAL TRIAL: NCT06935331
Title: Comparison of Opioid-Free Versus Traditional Opioid-Containing Postoperative Pain Management Pathways for Adolescent Idiopathic Scoliosis
Brief Title: Prospective Opioid-Free AIS Fusion
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9209
Record Dates: First submitted 2025-03-31; First posted 2025-04-20 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS)
Keywords: Adolescent Idiopathic Scoliosis (AIS); Opioid; Pain Management Pathway

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid-Free/Opioid-Avoidant (Experimental): Managed post-operatively with an opioid-free pain regimen which will include:
  Intrafascial injection of clonidine, epinephrine, ropivacaine, and toradol solution, diluted to 100mL and injected during closure of wound.
  Gabapentin PO 300 mg TID x 30 days.
  Toradol IV dosed per body weight, max 30 mg q 6 hours for 24-28 hours.
  Ibuprofen PO dosed per body weight q 6-8 hours once toradol discontinued and discharged home with PO tabs.
  Acetaminophen PO dosed per body weight and discharged home with PO tabs.
  Diazepam PO dosed per body weight during stay and discharged home with PO tabs.
  Non-medicinal therapy: Ice, Aromatherapy, Music therapy, Pet therapy, Early mobilization and PT.
  Interventions: Drug: Opioid-Free/Opioid-Avoidant
- Opioid-Containing (Active Comparator): Managed post-operatively with a traditional opioid containing pain regimen including:
  Intrafascial injection of clonidine, epinephrine, ropivacaine, and toradol solution, diluted to 100mL and injected during closure of wound.
  Post-operative morphine IV for breakthrough pain.
  Oral narcotic (hydrocodone/acetaminophen).
  Gabapentin PO 300 mg TID x 30 days.
  Toradol IV dosed per body weight, max 30 mg q 6 hours for 24-28 hours.
  Ibuprofen PO dosed per body weight q 6-8 hours once toradol discontinued and discharged home with PO tabs.
  Acetaminophen PO dosed per body weight and discharged home with PO tabs.
  Diazepam PO dosed per body weight during stay and discharged home with PO tabs.
  Non-medicinal therapy: Ice, Early mobilization and PT.
  Interventions: Drug: Opioid-Containing

INTERVENTIONS:
Drug: Opioid-Free/Opioid-Avoidant — Managed post-operatively with an opioid-free pain regimen which will include:
  Intrafascial injection of clonidine, epinephrine, ropivacaine, and toradol solution, diluted to 100mL and injected during closure of wound
  Gabapentin PO 300 mg TID x 30 days
  Toradol IV dosed per body weight, max 30 mg q 6 hours for 24-28 hours
  Ibuprofen PO dosed per body weight q 6-8 hours once toradol discontinued and discharged home with PO tabs
  Acetaminophen PO dosed per body weight and discharged home with PO tabs
  Diazepam PO dosed per body weight during stay and discharged home with PO tabs
  Non-medicinal therapy: Ice, Aromatherapy, Music therapy, Pet therapy, Early mobilization and PT
  Arms: Opioid-Free/Opioid-Avoidant
Drug: Opioid-Containing — Managed post-operatively with a traditional opioid containing pain regimen including:
  Intrafascial injection of clonidine, epinephrine, ropivacaine, and toradol solution, diluted to 100mL and injected during closure of wound
  Post-operative morphine IV for breakthrough pain
  Oral narcotic (hydrocodone/acetaminophen)
  Gabapentin PO 300 mg TID x 30 days
  Toradol IV dosed per body weight, max 30 mg q 6 hours for 24-28 hours
  Ibuprofen PO dosed per body weight q 6-8 hours once toradol discontinued and discharged home with PO tabs
  Acetaminophen PO dosed per body weight and discharged home with PO tabs
  Diazepam PO dosed per body weight during stay and discharged home with PO tabs
  Non-medicinal therapy: Ice, Early mobilization and PT
  Arms: Opioid-Containing

SUMMARY:
The purpose of this study is to compare the efficacy of a multimodal opioid-free (OF) pain management protocol with a traditional opioid-containing (OC) protocol in pediatric patients undergoing instrumented PSF for idiopathic scoliosis.

DETAILED DESCRIPTION:
Opioids are the most common controlled medication used medically and non-medically by adolescents in the United States. Opioid prescribing practices are inextricably linked with the ongoing public health crisis of opioid misuse in the peri-adolescent population. However, the immediate postoperative period following instrumented posterior spinal fusion (PSF) for idiopathic scoliosis represents a difficult challenge for patients and surgeons alike - particularly with regard to pain control. Opioid medications are commonly used to manage early postoperative pain in these patients, though are associated with potentially deleterious effects and remain at the center of a national health crisis. In particular for peri-adolescent patients, opioids are known to disrupt central nervous system maturation, which may lead to long-term behavioral dysfunction, including increased vulnerability to addiction in adulthood. On the other hand, it is well-recognized that inadequate pain control is associated with atelectasis, delayed mobilization, protracted hospitalization, and increased complication rates following posterior instrumented PSF for idiopathic scoliosis. Consequently, there is a rising, unmet need to develop postoperative recovery pathways for this population, aimed at efficient and safe pain management that minimizes or eliminates opioids while ensuring a positive postoperative experience for the patient.

Previous studies in adult and pediatric patients have compared traditional opioid-based pain regimens to opioid-sparing regimens in the perioperative period, but have been limited by high rates of crossover, retrospective designs, reliance on indwelling pain catheters, reliance on opioids for early postoperative analgesia, and/or lack of patient-reported outcomes. While there are growing efforts to investigate and adopt opioid-free (OF) protocols in adult orthopaedic patients, such protocols have yet to be thoroughly evaluated in the pediatric population. A prior study approved and completed (Protocol# PED032) by Dr. Michael Paloski and team demonstrated that a comprehensive, multimodal, OF pain management pathway following instrumented PSF for idiopathic scoliosis results in equivalent length of stay and fewer opioids prescribed at discharge compared with a traditional opioid-containing (OC) pathway. To our knowledge, this was the first study to show that completely OF postoperative pain management is possible in this population. Additional studies, including the study proposed here, are necessary to evaluate patient-reported outcomes in this population when OF pain management is utilized and to delineate patient-specific and procedure-specific details that may predict success with an OF regimen.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (10-20 years of age at the time of surgery)
* Diagnosis of idiopathic scoliosis
* Undergoing primary instrumented PSF

Exclusion Criteria:

* Age <10 years or >20 years at time of surgery
* Patients with non-idiopathic scoliosis etiology, ie neuromuscular or syndromic scoliosis
* Patients undergoing non-fusion spinal surgeries, ie growing rods or tethering

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain rating on the 10-point numeric pain rating scale (NPRS) | 24 hours after surgery completion
  Pain rating on the 10-point numeric pain rating scale (NPRS) 24 hours after surgery completion

SECONDARY OUTCOMES:
Morphine milliequivalents (MME) | Perioperative/Periprocedural
  Morphine milliequivalents (MME) while inpatient
Length of hospital stay | Perioperative/Periprocedural
  Length of hospital stay (in days/hours)
opioid medication prescribed | Perioperative/Periprocedural
  Presence of opioid medication prescribed at discharge
Clinic phone calls regarding uncontrolled pain | Through study completion, an average of 1 year
  Clinic phone calls regarding uncontrolled pain
Delayed opioid prescriptions sent | Through study completion, an average of 1 year
  Delayed opioid prescriptions sent
Opioid refills requested or sent | Through study completion, an average of 1 year
  Number of opioid refills requested or sent
Unplanned emergency department or clinic visits for pain | Through study completion, an average of 1 year
  Instances of unplanned emergency department or clinic visits for pain
Days missed from school | Through study completion, an average of 1 year
  Number of days missed from school
symptomatic pseudoarthrosis | Through study completion, an average of 1 year
  Incidence of symptomatic pseudoarthrosis, confirmed either with computed tomography or during subsequent surgery
Numeric Pain Rating Scale (NPRS) - Patient | Through study completion, an average of 1 year
  Numeric Pain Rating Scale (NPRS) according to the patient.
Perceived Numeric Pain Rating Scale (NPRS) - Parent/Guardian | Through study completion, an average of 1 year
  Perceived Numeric Pain Rating Scale (NPRS) according to Parent/Guardian (0-10 with 10 being the worst)
Patient Acceptable Symptom State (PASS) (patient) | Through study completion, an average of 1 year
  Patient Acceptable Symptom State (PASS) completed by patient, a single yes or no question
Patient Acceptable Symptom State (PASS) (parent/guardian) | Through study completion, an average of 1 year
  Patient Acceptable Symptom State (PASS) according to the parent/guardian, a single yes or no question
Opioid medication utilization | Through study completion, an average of 1 year
  Opioid medication utilization (Yes/No) after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Michael Paloski, DO, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (1):
- OrthoCarolina Research Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plan